CLINICAL TRIAL: NCT02479477
Title: Impact of Labour Kinesiotherapy in the Quality Life of Auxiliary Nursing in the Surgery Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Vera Lucia dos Santos Alves, Professor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14076613.0.0000.5479
Record Dates: First submitted 2015-06-18; First posted 2015-06-24 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Quality of Life; Pain
Keywords: Public Health; Nursing Staff, Hospital
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- kinesio therapy (Experimental): The intervention is one protocol of labour kinesiotherapy that will be realized tree times per week, eatch intervention with fiveteen minutes, during eitgh weeks.
  To change to sf-36 questionary after intervention. the intervention is the use of labour kinesio terapy in the auxiliary nursing The chance is in the score of questionary, the investigators hope that after intervention the score will increase.
  Interventions: Other: kinesio therapy
- control (No Intervention): the control group will continue their daily tasks uring eitgh weeks. To change to sf-36 questionary after intervention. the intervention is the use of labour kinesio terapy in the auxiliary nursing The chance is in the score of questionary, the investigators hope that after intervention the score will increase.

INTERVENTIONS:
Other: kinesio therapy — during for fifteen minutes the nursing assistants will perform stretching exercises and muscle relaxation of large muscle groups the orthostatic position
  Arms: kinesio therapy

SUMMARY:
The quality of life and daily activities can be affected by muscleskeletal pain and one of the forms of assessment is through the SF-36 questionnaire. The investigators know that the working kinesitherapy is a way to improve the quality of life.

DETAILED DESCRIPTION:
The activities in the work routine can cause pain and negatively affect quality of life. There is the hypothesis that gymnastics may be used for pain and injuries relating to repetitive movement at work. Objective the study is assess the impact of labor kinesiotherapy in the quality of life of the operating room nursing assistants.

ELIGIBILITY:
Inclusion Criteria:

* professional nursing assistants allocated in the surgical center at least one year
* both genders
* who agreed to participate in the study by signing the informed consent

Exclusion Criteria:

* persons submitted on any surgery in the last six months
* with illness or muscle-skeletal disabilities
* or who couldn't attend all sessions for vacations or scale

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change in questionnaire score after the intervention (minimum 0, maximum 100) | two months
  SF-36 domains